CLINICAL TRIAL: NCT04475354
Title: Mechanisms Explaining Psychological Distress In CErvical Cancer Patients and Partners (DICE): a Population-based Prospective Study
Brief Title: Distress In CErvical Cancer Patients and Partners
Acronym: DICE
Status: Recruiting | Type: Observational
Sponsor: Comprehensive Cancer Centre The Netherlands (Other)
Collaborators: Tilburg University (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Nicole Ezendam, Principal Investigator, Comprehensive Cancer Centre The Netherlands
Other Study IDs: NL.67509.028.18
Record Dates: First submitted 2020-01-16; First posted 2020-07-17 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cervical Cancer; Psychologic Stress; Psychological Distress; Survivorship; Quality of Life
MeSH Terms: conditions — Uterine Cervical Neoplasms; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: pro-and anti-inflammatory cytokines, telomere length Scalp hair: cortisol, melatonin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical cancer patients and their partners: 520 cervical cancer patients will complete questionnaires, online food diary and wear a fitbit after diagnosis, after 6 months, and after 1, 2, 5 and 10 years. In addition, a subsample (n=116) will donate blood samples and a scalp hair sample after diagnosis and 6, 12 and 24 months. We expect 312 partners of cervical cancer patients to included in the study and complete questionnaires after diagnosis, after 6 months, and after 1, 2, 5 and 10 years

SUMMARY:
Rationale: A growing number of cervical cancer patients live years beyond their cancer diagnosis and ultimately survive their disease. Cervical cancer patients report higher levels of psychological distress compared to other (gynecological) cancer types, resulting in physical and psychosocial limitations. The mechanisms explaining why some patients do, and others do not experience persistent psychological distress after cervical cancer remain unclear.

Objective: Gain insight into the mechanisms explaining psychological distress (i.e. anxiety, depression, cancer worry, perceived stress) in a prospective population-based sample of cervical cancer patients. Factors to be studied include characteristics of the individual (demographical and clinical, including comorbidities), characteristics of the environment ((sexual) relationships), biological function (cortisol, melatonin and sex hormone production assessed in scalp hair, inflammation and telomere length assessed in blood, overall quality of life (EORTC QLQ-C30), symptoms (EORTC QLQ-CX24), functional status (physical activity and sleep measured using the Actigraph activity tracker, and food intake measured using the online 'Eetmeter'), and general health perceptions (B-IPQ). The second aim is to assess the impact of cervical cancer on partners' distress (cancer worry, illness perceptions, relationship quality, dyadic coping).

DETAILED DESCRIPTION:
Study design: Prospective population-based study in which cervical cancer patients and their partners are included shortly after diagnosis and followed until 10 years after diagnosis. Patients from treatment centres in the Netherlands and their partners will be asked to complete questionnaires after diagnosis, after 6 months, and after 1, 2, 5 and 10 year. Clinical data like disease stage, initial treatment and mortality will be extracted from the Netherlands Cancer Registry. In a subsample of patients, additionally objective lifestyle (actigraph, biosensor) and biological (blood, hair) measures are assessed at diagnosis and after 6, 12 and 24 months. .

Study population: Newly diagnosed stage 1-3 cervical cancer patients (N=520) and their partners (N=312, expected) from any treatment centre in the Netherlands will be asked to fill out questionnaires. In a subsample of patients (N=116) additionally lifestyle and biological measures are assessed at all time-points.

Main study parameters/endpoints: psychological distress (anxiety, depression, perceived stress, cancer worry)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients and partners are asked to complete a questionnaire at 6 points in time: after diagnosis, after 6 months, and after 1, 2, 5 and 10 year. Patients will additionally be asked to complete an online food diary for 3 days. A subsample of patients will be asked to donate blood samples (2X10 ml, 10 minutes) to assess inflammation markers and telomere length, to donate a scalp hair sample (10 mg) to assess hormone production after diagnosis and after 6, 12 and 24 months, and to wear an Actigraph activity tracker to assess physical activity and sleep and a Philips Biosensor to assess heart rate variability as a marker of vagal nerve function at 6, 12 and 24 months.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Newly diagnosed with cervical cancer stage I, II or III
* >18 years or older

Exclusion Criteria:

* Participants with cognitive impairment will not be included because of expected difficulties in completing the questionnaires without assistance.
* Participants who are not able to read or write Dutch will be excluded, as they are not able to complete a Dutch questionnaire.

Partners

Inclusion Criteria:

* Partner of patient participating in the study
* >18 years

Exclusion Criteria:

* Participants with cognitive impairment will not be included because of expected difficulties in completing the questionnaires without assistance.
* Participants who are not able to read or write Dutch will be excluded, as they are not able to complete a Dutch questionnaire.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed I-III stage cervical cancer patients that receive primary treatment in one of the treatment centres will be identified by their treating gynaecologist. Patients will be invited before the start of treatment and will be followed until 10 years after diagnosis. Additionally, patients will be asked to invite their partner to participate.
Sampling Method: Probability Sample
Enrollment: 832 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety/ depression | 24 months
  Hospital Anxiety and Depression Scale (1-21, higher scores indicate more anxiety or depression)

SECONDARY OUTCOMES:
Cancer worry | 24 months
  Impact of Cancer version 2 (Worry Scale) (0-5, higher scores indicate more worry)
Perceived stress | 24 months
  Perceived Stress Scale (0-40, higher scores indicate more perceived stress)
Health-related quality of life | 24 months
  EORTC Quality of Life Questionnaire (QLQC30) (0-100, higher scores indicate better quality of life or more symptoms)
Cervical cancer health-related quality of life | 24 months
  EORTC Cervical Cancer Module (CX24) (0-100, higher scores indicate better quality of life or more symptoms)
Sexual Health | 24 months
  EORTC Sexual Health Questionnaire (SHQ22) (0-100, higher scores indicate better quality of life or more symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ezendam, Principal Investigator — Netherlands Comprehensive Cancer Organisation
Locations (6):
- Netherlands (6):
  - Amphia, Breda
  - Catharina Hospital, Eindhoven
  - University Medical Center Groningen, Groningen
  - MUMC, Maastricht
  - RadboudUMC, Nijmegen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Questionnaire data will be dissiminated 1 year after conclusion of the study. Data from the PROFILES registry are freely available for non-commercial scientific research, subject to study question, privacy and confidentiality restrictions, and registration (www.profileregistry.nl).

REFERENCES:
- See also: https://www.nvog.nl/organisatie/pijler-oncologie/dgog/studies/dice-2/ — https://www.profilesregistry.nl/